CLINICAL TRIAL: NCT05089539
Title: The Effect of Angiotensin Receptor-Neprilysin Inhibition on Cardiac Fibrosis in Patients With HFpEF: A Randomized Controlled Trial
Brief Title: The Effect of Angiotensin Receptor-Neprilysin Inhibition on Cardiac Fibrosis in Patients With HFpEF
Acronym: ARNICFH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, PhD, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-10-21
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFpEF with ARNI treatment (Experimental): Sacubitril/valsartan (ARNI, 100mg bid)
  Interventions: Drug: Angiotensin Receptor-Neprilysin Inhibition
- Control group (Placebo Comparator): placebo (100mg bid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Angiotensin Receptor-Neprilysin Inhibition — Sacubitril/valsartan [100 mg] bid). Continuous treatment was maintained for at least three months.
  Other Names: Sacubitril/valsartan
  Arms: HFpEF with ARNI treatment
Drug: Placebo — Placebo [100 mg] bid). Continuous treatment was maintained for at least three months.
  Arms: Control group

SUMMARY:
The effectively therapeutic approaches for Heart failure with preserved ejection fraction (HFpEF) remain limited. The PARAGON-HF trial found that Angiotensin Receptor-Neprilysin Inhibition (ARNI) has potential benefits for the management of HFpEF. Nevertheless, the role of ARNI in cardiac fibrosis in HFpEF are still unclear. We will conduct a prospective randomized controlled trial to evaluate the effect of ARNI on cardiac fibrosis in patients with HFpEF by cardiac magnetic resonance (CMR).

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) comprises approximately 50% of all heart failure. The effectively therapeutic approaches for HFpEF remain limited. The PARAGON-HF trial found that Angiotensin Receptor-Neprilysin Inhibition (ARNI) has potential benefits for the management of HFpEF. Nevertheless, the role of ARNI in cardiac fibrosis in HFpEF are still unclear. We will conduct a prospective randomized controlled trial to evaluate the effect of ARNI on cardiac fibrosis in patients with HFpEF by cardiac magnetic resonance (CMR). We will randomly assign 60 patients with HFpEF (NYHA II-IV) class, ejection fraction ≥ 50% and elevated level of natriuretic peptides to receive sacubitril-valsartan (target 100mg bid) or placebo (100mg bid). The primary endpoint is change in extracellular volume [ECV] measured by CMR. The secondary endpoints were 6-minute walking distance(6-WMD), KCCQ, hospitalizations for heart failure, myocardial infarction and death.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Age ≥ 45 years at time of screening
* Preserved systolic left ventricular function, defined by left ventricular ejection fraction (LVEF) ≥ 50%
* NYHA classes II-IV
* H2FPEF score ≥ 6 or HFA-PEFF score ≥ 5

Exclusion Criteria:

* Patients with a known history of angioedema
* History of hypersensitivity to ARNI
* Any prior echocardiographic measurement of LVEF <45%
* Significant congenital heart disease
* Rheumatic valvular heart disease
* Acute coronary syndrome, cardiac surgery, other major cardiovascular surgery
* Probable alternative diagnoses could account for the patient's HF symptoms
* Systolic blood pressure(BP) >180 mm Hg or diastolic BP >120 mm Hg at visit
* Diastolic BP <90 mm Hg at visit 1, or symptomatic hypotension
* Patients with a cardiac pacemaker therapy device
* eGFR <30 ml/min/1.73 m2
* Serum potassium >5.2 mmol/l at visit 1
* Pregnant or nursing women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular volume [ECV] | Before ARNI or placebo treatment and after 3 months of continuous ANRI or palcebo treatment
  Extracellular volume [ECV] assessment by CMR

SECONDARY OUTCOMES:
myocardial infarction, hospitalization for heart failure and death | After 3 months of continuous ANRI or palcebo treatment
  myocardial infarction, hospitalization for heart failure and all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Background] Vaduganathan M, Jhund PS, Claggett BL, Packer M, Widimsky J, Seferovic P, Rizkala A, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. A putative placebo analysis of the effects of sacubitril/valsartan in heart failure across the full range of ejection fraction. Eur Heart J. 2020 Jul 1;41(25):2356-2362. doi: 10.1093/eurheartj/ehaa184. PMID 32221596
- [Background] van der Meer P, Gaggin HK, Dec GW. ACC/AHA Versus ESC Guidelines on Heart Failure: JACC Guideline Comparison. J Am Coll Cardiol. 2019 Jun 4;73(21):2756-2768. doi: 10.1016/j.jacc.2019.03.478. PMID 31146820